CLINICAL TRIAL: NCT02162485
Title: Pharmacokinetic Study Comparing Salmeterol/Fluticasone Easyhaler Products and Seretide Diskus 50/500 µG/Inhalation; A Randomised, Open, Single Centre, Single Dose, Crossover Study in Healthy Subjects
Brief Title: Pharmacokinetic Study Comparing Salmeterol/Fluticasone Easyhaler Products and Seretide Diskus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3106009
Record Dates: First submitted 2014-06-05; First posted 2014-06-12 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate; Charcoal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Salmeterol/fluticasone Easyhaler (Experimental): Single dose of Salmeterol/fluticasone Easyhaler
  Interventions: Drug: Salmeterol/fluticasone Easyhaler
- Salmeterol/fluticasone Easyhaler with charcoal (Experimental): Single dose of Salmeterol/fluticasone Easyhaler with concomitant charcoal administration (Carbomix granules)
  Interventions: Drug: Salmeterol/fluticasone Easyhaler with charcoal
- Seretide Diskus (Active Comparator): Single dose of Seretide Diskus
  Interventions: Drug: Seretide Diskus
- Seretide Diskus with charcoal (Active Comparator): Single dose of Seretide Diskus with concomitant charcoal administration (Carbomix granules)
  Interventions: Drug: Seretide Diskus with charcoal

INTERVENTIONS:
Drug: Salmeterol/fluticasone Easyhaler
  Arms: Salmeterol/fluticasone Easyhaler
Drug: Salmeterol/fluticasone Easyhaler with charcoal
  Arms: Salmeterol/fluticasone Easyhaler with charcoal
Drug: Seretide Diskus
  Arms: Seretide Diskus
Drug: Seretide Diskus with charcoal
  Arms: Seretide Diskus with charcoal

SUMMARY:
The purposes of this study is to compare the test products Salmeterol/fluticasone Easyhaler with marketed product Seretide Diskus in terms of the drug absorbed into the blood stream

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained
* Good general health ascertained by detailed medical history, and laboratory and physical examinations

Exclusion Criteria:

* Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, GI, pulmonary, metabolic-endocrine, neurological or psychiatric disease within the previous 2 years
* Any condition requiring regular concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study. As an exception, paracetamol and ibuprofen for occasional pain are allowed
* Known hypersensitivity to the active substance(s) or the excipient (lactose, which contains small amounts of milk protein) of the drug
* Pregnant or lactating females

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Cmax of plasma salmeterol and fluticasone propionate | within 34 h
AUCt of plasma salmeterol and fluticasone propionate | 34 h

CONTACTS AND LOCATIONS:
Overall Officials: Merja Mäkitalo, Study Director — Orion Corporation, Orion Pharma; Leena Mattila, MD, PhD, Principal Investigator — Orion Pharma Clinical Pharmacology Unit, Espoo, Finland
Locations (1):
- Orion Pharma Pharmacology Unit, Espoo, Finland